CLINICAL TRIAL: NCT00005585
Title: ALINC #17 Treatment for Patients With Low Risk Acute Lymphoblastic Leukemia: A Pediatric Oncology Group Phase III Study
Brief Title: Combination Chemotherapy in Treating Children With Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9904; COG-P9904 (Other: Children's Oncology Group); POG-9904 (Other: Pediatric Oncology Group); CDR0000067657 (Other: Clinical Trials.gov); NCI-2012-02321 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2013-06

CONDITIONS: Leukemia
Keywords: childhood acute lymphoblastic leukemia in remission; B-cell childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia | interventions — Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Leucovorin; Mercaptopurine; Methotrexate; pegaspargase; Asparaginase; Thioguanine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm I: (combination chemotherapy) (Experimental): CONSOLIDATION: Pts receive Methotrexate(MTX) IV over 24 hrs on day 1 and oral leucovorin calcium (CF) every 6 hrs for 3 doses at 42 hours after initiation of MTX infusion during weeks 7, 10, 13, 16, and 19. Pts also receive MTX IT on wks 7, 10, 13, 16, 19, and 22; oral mercaptopurine(6-MP) daily wks 5-24; oral dexamethasone (DM) 2x on days 1-7 of wks 8 and 17; and vincristine sulfate (VCR) IV on day 1 of wks 8, 9, 17, and 18. CONTINUATION: Pts receive oral 6-MP daily on wks 25-130; oral DM twice a day on days 1-7 and vincristine sulfate (VCR) IV on days 1 and 8 during wks 25, 41, 57, 73, 89, and 105; oral MTX on wks 25-130 (except during wks of IT MTX); and MTX IT on wks 25, 37, 49, 61, 73, 85, 97, and 109.
  Interventions: Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: vincristine sulfate
- Arm II (combination chemotherapy) (Experimental): CONSOLIDATION: Pts receive methotrexate (MTX) IV over 4 hrs on day 1 and oral leucovorin calcium (CF) during wks 7, 10, 13, 16, and 19. Pts also receive MTX IT on wks 7, 10, 13, 16, 19, and 22; oral mercaptopurine (6-MP) daily on wks 5-24; oral dexamethasone (DM) 2x on days 1-7 of wks 8 and 17; and vincristine sulfate (VCR) IV on day 1 of wks 8, 9, 17, and 18. CONTINUATION: Pts receive oral 6-MP daily on wks 25-130; oral DM 2x on days 1-7 and vincristine sulfate (VCR) IV on days 1 and 8 during wks 25, 41, 57, 73, 89, and 105; oral MTX weekly on wks 25-130 (except during wks of IT MTX); and MTX IT on wks 25, 37, 49, 61, 73, 85, 97, and 109.
  Interventions: Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: vincristine sulfate
- Arm III (combination chemotherapy) (Experimental): CONSOLIDATION: Pts receive methotrexate (MTX) IV and leucovorin calcium (CF) as in arm I on wks 7, 10, 13, 24, 27, and 30. Pts also receive oral mercaptopurine (6-MP) daily on wks 5-13 and then on wk 24 and continuing until the end of consolidation; MTX IT on wks 7, 10, 13, 16, 20, 21, and 30; oral dexamethasone (DM) twice daily on days 1-7 of wks 8, 16-18, and 28; vincristine sulfate (VCR) IV on day 1 of wks 8, 9, 16-18, 28, and 29; pegaspargase intramuscularly on wk 16; daunorubicin hydrochloride IV on day 1 of wks 16-18; cyclophosphamide IV on day 1 of wk 20; cytarabine IV or subcutaneously on days 2-5 of wks 20 and 21; and oral thioguanine daily on days 1-14 of wks 20 and 21. CONTINUATION: Pts receive oral 6-MP daily on wks 33-130; oral dexamethasone (DM) twice a day on days 1-7 and VCR IV on days 1 and 8 during wks 41, 57, 73, 89, and 105; oral MTX weekly on wks 33-130 (except during wks of IT MTX); and MTX IT on wks 37, 49, 61, 73, 85, 97, and 109.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate
- .Arm IV (combination chemotherapy) (Experimental): CONSOLIDATION: Pts receive methotrexate (MTX) and leucovorin calcium (CF) on wks 7, 10, 13, 24, 27, and 30. Pts receive mercaptopurine(6-MP) daily weeks 5-13 then beginning wk 24 and continuing until end of consolidation; MTX on wks 7, 10, 13, 16, 20, 21, and 30; dexamethasone (DM) 2x daily on days 1-7 of wks 8, 16-18, and 28; vincristine sulfate (VCR) day 1 of wks 8, 9, 16-18, 28, and 29; pegaspargase on wk 16; daunorubicin hydrochloride on day 1 of wks 16-18; cyclophosphamide on day 1 of wk 20; cytarabine on days 2-5 of wks 20 and 21; thioguanine daily on days 1-14 of wks 20 and 21. CONTINUATION: Pts receive mercaptopurine(6-MP) daily on weeks 33-130; oral dexamethasone (DM) twice a day on days 1-7 and VCR IV on days 1 and 8 during weeks 41, 57, 73, 89, and 105; oral MTX weekly on weeks 33-130 (except during weeks of IV MTX); and IV MTX on weeks 37, 49, 61, 73, 85, 97, and 109.
  Interventions: Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: thioguanine; Drug: vincristine sulfate

INTERVENTIONS:
Drug: cyclophosphamide — Given IV
  Other Names: Cytoxan; NSC #26271
  Arms: .Arm IV (combination chemotherapy); Arm III (combination chemotherapy)
Drug: cytarabine — Deoxycytidine analogue which is metabolized to ARA-CTP, a substance which inhibits DNA polymerase.
  Other Names: cytosine arabinoside; Ara-C; Cytosar; NSC #063878
  Arms: .Arm IV (combination chemotherapy); Arm III (combination chemotherapy)
Drug: daunorubicin hydrochloride — Given IV
  Other Names: Daunomycin; rubidomycin; Cerubidine; NSC #82151
  Arms: .Arm IV (combination chemotherapy); Arm III (combination chemotherapy)
Drug: dexamethasone — Dexamethasone is a synthetic fluorinated glucocorticoid devoid of mineralocorticoid effects.
  Other Names: Decadron; NSC#034521
Drug: leucovorin calcium — Synthetic d,l-5 CHO tetrahydrofolate, which is used to bypass the inhibition of dihydrofolate reductase by Methotrexate (MTX)
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC#003590
Drug: mercaptopurine — An analogue of the nucleic acid constituent adenine and the physiological purine base hypoxanthine
  Other Names: 6-MP; Purinethol; NSC #00075
Drug: methotrexate — A folate analogue which inhibits the enzyme dihydrofolate reductase, haltin g DNA, RNA, and protein synthesis
  Other Names: MTX; amethopterin; NSC#00740; IND#4291
Drug: pegaspargase — E-Coli asparaginase deaminates asparagine, thus, is lethal for cells which cannot synthesize asparagine.
  Other Names: E Coli; Elspar; asparaginase; Erwinia; PEG; NSC#109229
  Arms: .Arm IV (combination chemotherapy); Arm III (combination chemotherapy)
Drug: thioguanine — Given orally
  Other Names: 6-thioguanine; 2-amino-1; 7-dihydro-6H-purine-6-thione; WR-1141; Tabloid; Lanvis; NSC # 752
  Arms: .Arm IV (combination chemotherapy); Arm III (combination chemotherapy)
Drug: vincristine sulfate — Given IV
  Other Names: Oncovin; VCR; LCR; NSC #67574

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells. It is not yet known which regimen of combination chemotherapy is more effective for childhood acute lymphoblastic leukemia.

PURPOSE: This randomized phase III trial is comparing different regimens of combination chemotherapy to see how well they work in treating children with acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy and toxicity of short methotrexate infusion vs longer infusion in patients with low-risk acute lymphoblastic leukemia.
* Compare the efficacy of these regimens of methotrexate, with or without multidrug intensification, in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to genetics (stratum 1: trisomy 4/10 but not TEL/AML1 vs stratum 2: TEL/AML1 with or without trisomy 4/10).

All patients receive induction therapy (weeks 1-4) on another protocol (POG-9900).

Stratum 1

* Consolidation therapy begins on week 5. Patients are randomized to arm I or II.

  * Arm I: Patients receive methotrexate (MTX) IV over 24 hours on day 1 and oral leucovorin calcium (CF) every 6 hours for 3 doses beginning 42 hours after initiation of MTX infusion during weeks 7, 10, 13, 16, and 19.
  * Arm II: Patients receive MTX IV over 4 hours on day 1 and oral CF as in arm I during weeks 7, 10, 13, 16, and 19.
* Patients in arms I and II also receive MTX intrathecally (IT) on weeks 7, 10, 13, 16, 19, and 22; oral mercaptopurine (6-MP) daily on weeks 5-24; oral dexamethasone (DM) twice daily on days 1-7 of weeks 8 and 17; and vincristine (VCR) IV on day 1 of weeks 8, 9, 17, and 18.

Stratum 2

* Consolidation therapy begins on week 5 and delayed intensification therapy begins on week 16. Patients are randomized to delayed intensification or no delayed intensification. Patients randomized to no delayed intensification are then randomized to consolidation therapy on arm I or II. Patients randomized to delayed intensification are then randomized to arm III or IV. Patients with trisomy 4/10 are not randomized to arms III and IV.

  * Arm III: Patients receive MTX IV and CF as in arm I on weeks 7, 10, 13, 24, 27, and 30.
  * Arm IV: Patients receive MTX IV and CF as in arm II on weeks 7, 10, 13, 24, 27, and 30.
* Patients in arms III and IV also receive oral 6-MP daily on weeks 5-13 and then beginning on week 24 and continuing until the end of consolidation; MTX IT on weeks 7, 10, 13, 16, 20, 21, and 30; oral DM twice daily on days 1-7 of weeks 8, 16-18, and 28; VCR IV on day 1 of weeks 8, 9, 16-18, 28, and 29; pegaspargase intramuscularly on week 16; daunorubicin IV on day 1 of weeks 16-18; cyclophosphamide IV on day 1 of week 20; cytarabine IV or subcutaneously on days 2-5 of weeks 20 and 21; and oral thioguanine daily on days 1-14 of weeks 20 and 21.

All patients then receive continuation therapy beginning on week 25 for arms I and II and week 33 for arms III and IV and continuing until week 130 for all arms.

Continuation

* Arms I and II: Patients receive oral 6-MP daily on weeks 25-130; oral DM twice a day on days 1-7 and VCR IV on days 1 and 8 during weeks 25, 41, 57, 73, 89, and 105; oral MTX weekly on weeks 25-130 (except during weeks of IT MTX); and MTX IT on weeks 25, 37, 49, 61, 73, 85, 97, and 109.
* Arms III and IV: Patients receive oral 6-MP daily on weeks 33-130; oral DM twice a day on days 1-7 and VCR IV on days 1 and 8 during weeks 41, 57, 73, 89, and 105; oral MTX weekly on weeks 33-130 (except during weeks of IT MTX); and MTX IT on weeks 37, 49, 61, 73, 85, 97, and 109.

Patients are followed every 2 months for 2 years, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total 902 patients will be accrued for this study within 3.22 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell precursor acute lymphoblastic leukemia

  * Registered on POG-9900 Classification Study
* Registered within 7 days of documenting complete response (CR) after induction therapy on day 29 or, if 2 more weeks of induction are required, within 7 days of CR determination
* Classified as low-risk:

  * WBC less than 50,000/mm^3
  * Age 1 to 9
  * No adverse translocations [E2A-PBX1, t(1;19) or BCR/ABL, t(9;22); and MLL rearrangements]
  * No CNS 3 disease (CSF WBC at least 5/mm^3 with blasts present)
  * No testicular disease
  * At least one of the following present:

    * TEL/AML1, t(12;21)
    * Simultaneous trisomy of chromosomes 4 and 10

PATIENT CHARACTERISTICS:

Age:

* 1 to 9

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 838 (Actual)
Dates: Start 2000-04; Primary Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 4 years
  The test statistic will compare Kaplan-Meier curves with sample size derived from a modification of the Makuch-Simon method for historical controls
Occurrence of anticipated failures | Up to 7 years
  An O'Brien-Fleming analysis will be conducted, with significance declared if the observed logrank Z-statistic exceeds the z/sqrt(IF), where IF=fraction of anticipated failures that have occurred and z=critical value of the final analysis.
Grade 3 or greater CNS toxicity rates assessed using NCI CTC version 2.0 | Up to 7 years

SECONDARY OUTCOMES:
Measures of laboratory factors (other than MRD) | Up to 7 years
  Cox multiple regression will be utilized.
Homocysteine levels | Up to 7 years
  Will be correlated to acute neurotoxicity by Cox regression.

CONTACTS AND LOCATIONS:
Overall Officials: Paul L. Martin, MD, Study Chair — Duke Cancer Institute
Locations (123):
- United States (108):
  - Comprehensive Cancer Center at University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama Cancer Research Institute, Mobile, Alabama
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Stanford Cancer Center at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center/Kaiser Foundation Hospital - San Diego, San Diego, California
  - Children's Hospital and Health Center - San Diego, San Diego, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Broward General Medical Center, Fort Lauderdale, Florida
  - Children's Hospital of Southwest Florida, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Joe DiMaggio Children's Hospital at Memorial, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Clinic-Orlando, Orlando, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Scottish Rite Campus, Atlanta, Georgia
  - MBCCOP-Medical College of Georgia Cancer Center, Augusta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Rush University Medical Center, Chicago, Illinois
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Tulane Cancer Center at Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Children's Hospital of New Orleans, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Pediatric Specialty Clinic at Eastern Maine Medical Center, Bangor, Maine
  - Maine Children's Cancer Program, Scarborough, Maine
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed Army Medical Center, Silver Spring, Maryland
  - Floating Hospital for Children, Boston, Massachusetts
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - UMASS Memorial Cancer Center - University Campus, Worcester, Massachusetts
  - Children's Hospital of Michigan, Detroit, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Keesler Medical Center - Keesler Air Force Base, Keesler Air Force Base, Mississippi
  - University of Missouri - Columbia, Columbia, Missouri
  - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - St. Louis Children's Hospital, St Louis, Missouri
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Mount Sinai Medical Center, New York, New York
  - Beth Israel Medical Center - Singer Division, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Long Island Cancer Center at Stony Brook University Hospital, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Leo W. Jenkins Cancer Center at Pitt County Memorial Hospital, Greenville, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - Oklahoma University Medical Center, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Greenville Hospital System, Greenville, South Carolina
  - East Tennessee State University Cancer Center at Johnson City Medical Center, Johnson City, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Cancer Center at University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Children's Cancer Center and Hematology Service at Texas Children's Hospital, Houston, Texas
  - San Antonio Military Pediatric Cancer and Blood Disorders Center, Lackland Air Force Base, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - MBCCOP - South Texas Pediatrics, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Center for Cancer Prevention and Care at Scott and White Clinic, Temple, Texas
  - Vermont Cancer Center at University of Vermont, Burlington, Vermont
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - INOVA Fairfax Hospital, Falls Church, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Massey Cancer Center at Virginia Commonwealth University, Richmond, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Madigan Army Medical Center, Tacoma, Washington
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Clinic Research Foundation, Marshfield, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Australia (3):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - Royal Children's Hospital, Brisbane, Queensland
  - Royal Children's Hospital, Parkville, Victoria
- Canada (8):
  - Alberta Children's Hospital, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre de Recherche du Centre Hospitalier de l'Universite Laval, Sainte-Foy, Quebec
- University Medical Center Groningen, Groningen, Netherlands
- San Jorge Children's Hospital, Santurce, Puerto Rico
- Switzerland (2):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva

REFERENCES:
- [Background] Rabin KR, Gramatges MM, Borowitz MJ, Palla SL, Shi X, Margolin JF, Zweidler-McKay PA. Absolute lymphocyte counts refine minimal residual disease-based risk stratification in childhood acute lymphoblastic leukemia. Pediatr Blood Cancer. 2012 Sep;59(3):468-74. doi: 10.1002/pbc.23395. Epub 2011 Nov 18. PMID 22102553
- [Background] Xu H, Cheng C, Devidas M, Pei D, Fan Y, Yang W, Neale G, Scheet P, Burchard EG, Torgerson DG, Eng C, Dean M, Antillon F, Winick NJ, Martin PL, Willman CL, Camitta BM, Reaman GH, Carroll WL, Loh M, Evans WE, Pui CH, Hunger SP, Relling MV, Yang JJ. ARID5B genetic polymorphisms contribute to racial disparities in the incidence and treatment outcome of childhood acute lymphoblastic leukemia. J Clin Oncol. 2012 Mar 1;30(7):751-7. doi: 10.1200/JCO.2011.38.0345. Epub 2012 Jan 30. PMID 22291082
- [Background] Borowitz MJ, Devidas M, Hunger SP, et al.: Prognostic signficance of end consolidation minimal residual disease (MRD) in childhood acute lymphoblastic leukemia (ALL): A report from the Children's Oncology Group (COG). [Abstract] J Clin Oncol 26 (Suppl 15): A-10000, 2008.
- [Background] Borowitz MJ, Devidas M, Hunger SP, Bowman WP, Carroll AJ, Carroll WL, Linda S, Martin PL, Pullen DJ, Viswanatha D, Willman CL, Winick N, Camitta BM; Children's Oncology Group. Clinical significance of minimal residual disease in childhood acute lymphoblastic leukemia and its relationship to other prognostic factors: a Children's Oncology Group study. Blood. 2008 Jun 15;111(12):5477-85. doi: 10.1182/blood-2008-01-132837. Epub 2008 Apr 3. PMID 18388178
- [Background] Davies SM, Borowitz MJ, Rosner GL, Ritz K, Devidas M, Winick N, Martin PL, Bowman P, Elliott J, Willman C, Das S, Cook EH, Relling MV. Pharmacogenetics of minimal residual disease response in children with B-precursor acute lymphoblastic leukemia: a report from the Children's Oncology Group. Blood. 2008 Mar 15;111(6):2984-90. doi: 10.1182/blood-2007-09-114082. Epub 2008 Jan 8. PMID 18182569
- [Background] Hinds PS, Hockenberry MJ, Gattuso JS, Srivastava DK, Tong X, Jones H, West N, McCarthy KS, Sadeh A, Ash M, Fernandez C, Pui CH. Dexamethasone alters sleep and fatigue in pediatric patients with acute lymphoblastic leukemia. Cancer. 2007 Nov 15;110(10):2321-30. doi: 10.1002/cncr.23039. PMID 17926333
- [Background] Winick N, Martin PL, Devidas M, et al.: Delayed intensification (DI) enhances event-free survival (EFS) of children with B-precursor acute lymphoblastic leukemia (ALL) who received intensification therapy with six courses of intravenous methotrexate (MTX): POG 9904/9905: a Children's Oncology Group study (COG). [Abstract] Blood 110 (11): A-583, 2007.
- [Derived] Ramsey LB, Panetta JC, Smith C, Yang W, Fan Y, Winick NJ, Martin PL, Cheng C, Devidas M, Pui CH, Evans WE, Hunger SP, Loh M, Relling MV. Genome-wide study of methotrexate clearance replicates SLCO1B1. Blood. 2013 Feb 7;121(6):898-904. doi: 10.1182/blood-2012-08-452839. Epub 2012 Dec 11. PMID 23233662
- [Derived] Yang JJ, Cheng C, Devidas M, Cao X, Campana D, Yang W, Fan Y, Neale G, Cox N, Scheet P, Borowitz MJ, Winick NJ, Martin PL, Bowman WP, Camitta B, Reaman GH, Carroll WL, Willman CL, Hunger SP, Evans WE, Pui CH, Loh M, Relling MV. Genome-wide association study identifies germline polymorphisms associated with relapse of childhood acute lymphoblastic leukemia. Blood. 2012 Nov 15;120(20):4197-204. doi: 10.1182/blood-2012-07-440107. Epub 2012 Sep 24. PMID 23007406
- See also: Data Available: Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive — https://nctn-data-archive.nci.nih.gov/